CLINICAL TRIAL: NCT02170194
Title: GETSmart: Guided Education and Training Via Smart Phones to Promote Resilience
Acronym: GETSmart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 388404; 399461 (Other: Walter Reed National Military Medical Center)
Record Dates: First submitted 2014-06-09; First posted 2014-06-23 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Subthreshold PTSD
Keywords: smart phone apps; subthreshold PTSD; resilience enhancement; military veterans; natural disasters; terrorism; shootings; fMRI; physiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resilience Enhancement Group (Experimental): The resilience enhancement group will begin with a 90-minute session with the study psychologist, which will include a brief introduction to cognitive behavioral therapy (CBT), but focus primarily on psychoeducational, relaxation techniques and planning positive activities. The majority of the time will be focused on reviewing techniques that promote stress management. Emphasis will be placed on relaxation approaches such as controlled breathing, meditation and yoga. Focus will also be aimed at reviewing how engagement in positive activities may help prevent avoidance, promote social support and wellness. Over the subsequent 6 weeks, daily text messages to all participants will accentuate the positive, including providing recommendations on beneficial activities to engage in, encouraging such activities including in vivo exposure, and fostering behavioral changes.
  Interventions: Behavioral: Resilience Enhancement Training via Smart Phone
- Control Group (Placebo Comparator): The control group will be provided with an initial informational session providing them with details of where they can get help if they have worsened symptoms over time. In addition, the psychologist will briefly review the apps, but not provide the same pscyhoeducational detail given to the resilience enhancement group. They will receive daily texts with inspirational aphorisms (e.g., "Early to bed and early to rise makes a man healthy, wealthy, and wise.") for 6 weeks.
  Interventions: Behavioral: Daily Text Messages

INTERVENTIONS:
Behavioral: Resilience Enhancement Training via Smart Phone
  Arms: Resilience Enhancement Group
Behavioral: Daily Text Messages
  Arms: Control Group

SUMMARY:
There is no question that combat and domestic attacks can be stressful, and can have effects that last for months or even years, including reliving some of the events through nightmares or flashbacks, wanting to avoid anything that is a reminder of combat or domestic attack such as movies or the nightly news, or being jumpy and concerned about security. When someone has a lot of these symptoms they might be told they have PTSD, but even when that person doesn't have the full condition, just having some symptoms can affect their ability to function at the highest level at home, work, or in social settings, and puts you at greater risk for developing full PTSD. While someone who went through a significant stressful event might not need a long course of therapy if they don't have full PTSD, the investigator of this study thinks that working with them from a distance through their smart phone over time may decrease their symptoms, help them feel better, and prevent full PTSD. Thus the purpose of this study is to assess how a brief, relatively simple resiliency enhancement strategy, provided mostly through smart phones, affects someone with stress-related symptoms.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) has been identified in 10-20% of U.S. military service members (SMs) returning from Afghanistan and Iraq, and is associated with impaired physical health, mental health, and overall functional status. Resilience has often been spoken of, yet proven methods for promoting resilience, and protecting SMs from PTSD, have yet to be established. One easy and effective way of identifying those at higher risk for development of PTSD is through the one-page, 17-item self-administered PTSD Checklist (PCL). The total score can range from 17 to 85, and a score of 50 is the best cut-off for making a diagnosis of PTSD, but there are many military SMs who have impaired function associated with scores below this level. There have also been some high-profile fatal shootings on military installations in recent years, including Fort Hood, TX, and the Washington Naval Yard in the District of Columbia, and such incidents tend to be followed by persistent symptoms in many individuals who were in the vicinity at the time. There is limited recent evidence to suggest that lower intensity intervention might be effective in those with subthreshold PTSD, even though it does not necessarily successfully treat fully developed PTSD. We will therefore conduct a randomized controlled clinical trial involving 144 individuals who are eligible for care in the military healthcare system who report subthreshold PCL scores (28 to 49), either within five years after their return from Afghanistan or Iraq, or after being affected in some significant way by a terrifying incident such as a bombing or shooting, or a major natural disaster that results in significant loss of life such as a hurricane, tornado, or earthquake. Seventy-two participants will be assigned to the resilience enhancement group, which will be initiated with a single 90-minute introduction to both cognitive behavioral therapy (CBT) techniques and the use of smart-phone based applications (apps) that promote increased resilience through relaxation, biofeedback, psychoeducation and other techniques. Over the subsequent 6 weeks, daily text messages to all participants will accentuate the positive, including providing recommendations on beneficial activities, fostering behavioral changes, and in particular encouraging the completion of smart phone-based applications (apps). The control group (n=72) will be provided with an initial informational session providing them with details of where they can get help if they have worsened symptoms over time. They will receive daily texts with aphorisms for 6 weeks. Symptoms will be re-assessed with the PCL by personal computer (PC), tablet or smartphone based access to the NIH Clinical Trials Survey System (CTSS) for both the resilience enhancement and control groups at the end of each week in the 6-week training period. In addition the GAD, PHQ-9, and PCL will be assessed at baseline and 6weeks and at 3, 6 and 12 months. We anticipate that this relatively inexpensive resilience enhancement program will reduce the incidence of PTSD over the initial 6 weeks by 20% compared to the control group, and that this improvement will be maintained over the subsequent year. We further expect that the training program will be associated with a reduction in the incidence of PTSD by at least 10% over the follow-up period. Our power estimates indicate that with 72 participants each in the resilience enhancement and control groups, we will have 90% power to identify a significant difference between the two groups with 95% confidence (p < 0.05). For approximately 20% of participants (n=30; 15 in each group) we will perform psychophysiologic measures and functional MRI of the brain using the Affective Stroop paradigm at baseline and again 3-6 months later to assess for changes with resilience enhancement.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have had a deployment in Iraq or Afghanistan or exposure to a stressful event such as a domestic terrorist incident or natural disaster.
2. Participants must be in the United States and have an I-phone or Android platform smart phone and a service plan that includes the ability to receive text messages.
3. PTSD Checklist (PCL) score must be in the range of 28 to 49 at baseline.
4. No active suicidal ideation, as manifest by a response of "not at all" to the PHQ-9 question, "Over the past 2 weeks, how often have you been bothered by thoughts that you would be better off dead or of hurting yourself in some way?" .This will be assessed after written informed consent is attained.
5. No active PTSD diagnosis. This will be assessed by asking the participant and confirmed by the screening PCL and the baseline PCL.

   -

Exclusion Criteria:

All participants must adhere to the above inclusion criteria. However for those wishing to taking part in the on-site assessment, the following additional exclusion criteria will prevent them from taking part in the on-site fMRI and physiologic assessments, though they will still be able to take part in the GETSmart resilience enhancement vs. control groups:

1. Pregnancy: urine pregnancy tests will be performed on all females prior to the conduct of imaging studies both at baseline and follow-up assessments; women with positive tests upon baseline assessment will be excluded from the on-site assessment element; if a positive pregnancy test is identified at the follow up in-person assessment, the physiologic element will still be conducted but the MRI will not be performed.
2. Individuals with shrapnel, body piercings that cannot be removed, or other imbedded metal resulting from either trauma or surgical procedures will be excluded from the in-person assessments due to the risk or displacement of metal with magnetic resonance imaging;
3. Those with significant claustrophobia, including but not limited to intolerance of magnetic resonance imaging in the past, will be excluded from the in-person assessments, as we cannot provide sedating medications with the scans due to the potential impact of the medications on interpretation of scan results.
4. Individuals who are on calcium channel blockers (e.g., verapamil, nifedipine) or alpha blockers (e.g., prazosin, terazosin) who are unable to hold these medications for a 24-hour period prior to scanning, will be excluded from the in-person assessments due to the impact of these medications on the interpretation of fMRI imaging.
5. Those who are not eligible for care in the military healthcare system (DEERS-eligible) will be excluded from the in-person assessments.

   -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-05; Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist (PCL) | change from baseline at 6 weeks
  The PCL is a self-administered screen for PTSD (used both as a brief initial screen to confirm eligibility, and to provide a brief alternative in case some participants are unable to complete the more cumbersome CAPS at one or more follow-up intervals; demonstrates); a recent assessment of its psychometric properties in male veterans found very high internal consistency and convergent validity with the gold-standard CAPS (correlation, r=0.79). It should be noted that there is a military version of the PCL which we have used in prior studies that have involved solely military service members, the only difference between the military version and the more generalizable "civilian" version is the inclusion of the word "military" prior to "stressful experience" for 6 of the 17 items, so that there should not be a significant difference in the responses of service members who complete the civilian version, whereas the military version would not make sense for civilian participants
PTSD Checklist (PCL) | 3 months
  The PCL is a self-administered screen for PTSD (used both as a brief initial screen to confirm eligibility, and to provide a brief alternative in case some participants are unable to complete the more cumbersome CAPS at one or more follow-up intervals; demonstrates); a recent assessment of its psychometric properties in male veterans found very high internal consistency and convergent validity with the gold-standard CAPS (correlation, r=0.79). It should be noted that there is a military version of the PCL which we have used in prior studies that have involved solely military service members, the only difference between the military version and the more generalizable "civilian" version is the inclusion of the word "military" prior to "stressful experience" for 6 of the 17 items, so that there should not be a significant difference in the responses of service members who complete the civilian version, whereas the military version would not make sense for civilian participants
PTSD Checklist (PCL) | 6 months
  The PCL is a self-administered screen for PTSD (used both as a brief initial screen to confirm eligibility, and to provide a brief alternative in case some participants are unable to complete the more cumbersome CAPS at one or more follow-up intervals; demonstrates); a recent assessment of its psychometric properties in male veterans found very high internal consistency and convergent validity with the gold-standard CAPS (correlation, r=0.79). It should be noted that there is a military version of the PCL which we have used in prior studies that have involved solely military service members, the only difference between the military version and the more generalizable "civilian" version is the inclusion of the word "military" prior to "stressful experience" for 6 of the 17 items, so that there should not be a significant difference in the responses of service members who complete the civilian version, whereas the military version would not make sense for civilian participants
PTSD Checklist (PCL) | 12 months
  The PCL is a self-administered screen for PTSD (used both as a brief initial screen to confirm eligibility, and to provide a brief alternative in case some participants are unable to complete the more cumbersome CAPS at one or more follow-up intervals; demonstrates); a recent assessment of its psychometric properties in male veterans found very high internal consistency and convergent validity with the gold-standard CAPS (correlation, r=0.79). It should be noted that there is a military version of the PCL which we have used in prior studies that have involved solely military service members, the only difference between the military version and the more generalizable "civilian" version is the inclusion of the word "military" prior to "stressful experience" for 6 of the 17 items, so that there should not be a significant difference in the responses of service members who complete the civilian version, whereas the military version would not make sense for civilian participants

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ) | baseline, 6 weeks, 3 months, 6 months, 12 months
  The PHQ-9 is a brief screening instrument that is widely used to screen for and monitor the severity of depression. The GAD-7 provides similar validate efficacy in the screening and monitoring of anxiety spectrum disorders including generalized anxiety disorder, panic, social anxiety, and posttraumatic stress disorder. Both are elements of the PHQ, which was initially validated in 3000 primary care patients, including 500 at Walter Reed, where the PI of this protocol was the site PI.

OTHER OUTCOMES:
Functional magnetic resonance imaging (fMRI) | baseline, 3 months
  Functional magnetic resonance imaging (fMRI) is a potent, relatively novel method for objectively assessing the impact of posttraumatic stress disorder on the central nervous system. There are several variants of fMRI, but the most widely used, best studied method is known as BOLD (blood oxygen level dependent). Exposure to sensory stimuli results in neuronal activation in corresponding areas of the brain, which increases oxygen uptake in these areas. This results in a transient (3-6 seconds) decrease in blood oxygen levels in these areas, but there is a prompt response to increase blood flow to these areas, resulting in a more sustained increase in oxygenation which overwhelms the initial increase in extraction from these areas. T2-weighted images on fMRI show greater intensity in areas of increased oxygenation.
Psychophysiology | baseline, 3 months
  The Biopac recording software physiologic monitoring system that will measure heart rate (HR), heart rate variability (HRV), blood pressure (BP), respiratory rate (RR), and skin conductance (SC) at baseline, and throughout a fear conditioning task and Virtual Iraq sequences. The conditioning procedure will be used in which one of two conditioned stimuli (CS) will be paired with an aversive stimulus. Aversive stimuli will consist of airpuffs. There will be three phases: habituation, acquisition, and extinction. In the habituation phase, the CS will be presented without aversive stimuli. In the acquisition phase, the CS+ but not the CS- will be reinforced with an aversive stimulus. In the extinction phase, the two CS will not be reinforced.

CONTACTS AND LOCATIONS:
Locations (1):
- Uniformed Services University of the Health Sciences and Walter Reed National Military Medical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: Center for Neuroscience and Regenerative Medicine — http://braininjuryresearch.usuhs.edu/